CLINICAL TRIAL: NCT07067346
Title: A Study to Evaluate Safety and Efficacy of Radiopharmaceutical IR-101 in Patients With Relapsed or Refractory Neuroblastoma
Brief Title: Safety & Efficacy of IR-101 in Relapsed/Refractory Neuroblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Rong Tian, Director, Sichuan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HX2501
Record Dates: First submitted 2025-06-24; First posted 2025-07-16 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Neuroblastoma
Keywords: Radiopharmaceutical
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Study drug IR-101 Dose Escalation
  Interventions: Drug: IR-101

INTERVENTIONS:
Drug: IR-101 — IR-101 Dose Escalation

SUMMARY:
Radiopharmaceutical in Relapsed/Refractory Neuroblastoma

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory high-risk neuroblastoma with MIBG avid lesions in accordance with the Revised International Neuroblastoma Response Criteria (INRC);
2. All soft-tissue lesions detected on CT/MRI must be MIBG-avid;
3. Age ≥12 months;
4. Lansky performance status ≥50%;
5. Adequate organ function and hematologic parameters;

Exclusion Criteria:

1. Antibody-based immunotherapy within 5 half-lives or 30 days (whichever is shorter), or not yet recovered from adverse reactions of prior biologic therapies；
2. Treatment with [¹³¹I]MIBG or Lu-177 targeted radionuclide therapy <3 months of last administration;
3. Autologous transplant <12 weeks, or Allogeneic transplant <4 months (patients >4 months post-transplant must be free of active GVHD);
4. Radiotherapy within 2 weeks prior to first dose of study drug (However, if the subjects undergone radiotherapy for the sole lesion have MIBG uptake after 2 weeks of radiotherapy completion, they will be eligible); or Extensive-field radiotherapy (e.g., Cranio-spinal cord, whole lung, whole abdomen, or >50% bone marrow) within 12 weeks prior to first dose of study drug;
5. Renal Insufficiency;
6. Active Infections;

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of dose-limiting toxicities (DLTs) | From administration of IR-101 until 4 weeks after injection
  Incidence and severity of dose-limiting toxicities (DLTs)
Incidence and severity of adverse events (AEs) as assessed by CTCAE v5.0 | From administration of IR-101 until 4 weeks after last dose of injection
  Incidence and severity of adverse events (AEs) as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC) | 4 weeks after IR-101 administration
  Response assessed in accordance with the Revised International Neuroblastoma Response Criteria (INRC)
Absorbed radiation dose (Gy) distribution in normal organs and tumors by quantitative SPECT/CT dosimetry | About 21hours from time of IR-101 administration
  Absorbed radiation dose (Gy) distribution in normal organs and tumors by quantitative SPECT/CT dosimetry

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tian, MD, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - West China Hospital, Chengdu, Sichuang
  - West China Hospital, Chengdu

IPD SHARING:
Plan to Share IPD: No